CLINICAL TRIAL: NCT02735941
Title: Expression of G Protein-coupled Receptors and Ligands in Inflammatory Bowel Diseases and Colon Cancer
Brief Title: Study on Cannabinoid Receptor Expression in Gastrointestinal Diseases
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: KLI 521-B31
Record Dates: First submitted 2016-02-01; First posted 2016-04-13 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Colon Cancer
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, serum, biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- UC group: Patients with ulcerative colitis (active or remission)
- CD group: Patients with Crohn's disease (active or remission)
- Colon cancer group: Patients with colon cancer or metastasis
- control group: healthy individuals

SUMMARY:
The purpose of the study is to investigate phospholipid ligands and their receptors in inflammatory bowel diseases and colon cancer. Several new species of lipids have been recently discovered which are able to transmit information to cancer cells in the large intestine. The lipids and their responsive receptors build an axis that is thought to influence the development of inflammation and cancer.

DETAILED DESCRIPTION:
Expression of cannabinoid receptors are examined in mucosal biopsies of the colon and blood leukocytes of patients with inflammatory bowel disease (IBD) or colon cancer in comparison to healthy individuals by polymerase chain reaction, Western Blots and flow cytometry. Colonic endoscopic biopsies and blood are collected from adult patients with confirmed active Ulcerative colitis (UC) and Crohn's disease (CD), adult UC and CD patients in remission, colon cancer patients and from healthy individuals (controls). Biopsies from healthy individuals (control group) will have undergone colonoscopy during standard screening for colorectal cancer or for the diagnostic workup of gastrointestinal symptoms without endoscopic or histologic evidence of colonic disease. For UC patients, duration and location of disease (Montreal classification), endoscopic (Mayo score) and clinical activity score, histological features and current and previous treatments (5-aminosalicylic acid, corticosteroids, immunomodulators) will be recorded. For CD patients, duration and location of disease is assessed, a HarveyBradshaw Index and activity will be scored, histological features and current and previous treatments will be recorded. Blood is collected and immediately processed for flow cytometric experiments. Phospholipids are measured in serum and in colonic mucosal biopsy samples of all cohorts by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative colitis (active/remission)
* or Crohn's disease (active/remission)
* or Colon cancer (or metastasis)

Exclusion Criteria:

* unable to give informed consent
* pregnancy
* intermittent illness or comorbidity during Crohn/Ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing colon cancer screening program at the IBD outpatients clinic of the Medical University of Graz
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Analysis of cannabinoid receptors in blood leukocytes and biopsies from patients with IBD and colon cancer | within 24 months
  Protein content of cannabinoid receptors and G protein-coupled receptor 55 are measured by flow cytometry in blood leukocytes of patients with ulcerative colitis or Crohn's disease, and of healthy individuals. Transcripts of cannabinoid receptors and G protein-coupled receptor 55 are also measured in colonic mucosal biopsies of IBD/colon cancer patients and healthy individuals by polymerase chain reaction.

SECONDARY OUTCOMES:
Assessment of endoscopic activity scores (Mayo, Harvey Bradshaw index) in IBD patients. | within 24 months
Assessment of malignancy of colon cancer by tumor staging | within 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Schicho, PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No